CLINICAL TRIAL: NCT06942416
Title: Phase II, Single-Arm, Multicenter Clinical Study of Iparomlimab and Tuvonralimab in Combination With Paclitaxel Plus Cisplatin/Carboplatin and Radiotherapy for the Treatment of Locally Recurrent and Oligometastatic Cervical Cancer
Brief Title: Iparomlimab and Tuvonralimab With Chemoradiation for the Treatment of Locally Recurrent and Oligometastatic Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Peng Xie, Director, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2025-028-02
Record Dates: First submitted 2025-03-31; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Cervical Cancer; Neoplasm Recurrence, Local; Oligometastatic
Keywords: Immunotherapy; Paclitaxel; Cisplatin; Carboplatin; Radiation Therapy; Clinical Trials, Phase II as Topic; Progression-Free Survival; Biomarkers, Tumor; Treatment Outcome; Safety; Iparomlimab and Tuvonralimab
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasm Recurrence, Local; Neoplasms | interventions — Paclitaxel; Cisplatin; Carboplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chemotherapy+Immunotherapy+Radiotherapy (Experimental): Chemotherapy：TP (Paclitaxel and Cisplatin/Carboplatin); Immunotherapy：Iparomlimab and Tuvonralimab;Radiotherapy：All tumor lesions will be irradiated
  Interventions: Drug: Paclitaxel and Cisplatin/ Carboplatin; Drug: Iparomlimab and Tuvonralimab; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Paclitaxel and Cisplatin/ Carboplatin — Paclitaxel and Cisplatin Paclitaxel: 135 mg/m², intravenous infusion, Day 1, every 3 weeks (Q3W). Cisplatin: 75 mg/m², intravenous infusion, Days 1-3, every 3 weeks (Q3W). Carboplatin 0.3-0.4g/m², intravenous infusion, Day 1, Q3W .Duration: 4-6 cycles.
Drug: Iparomlimab and Tuvonralimab — Iparomlimab and Tuvonralimab 5mg/kg, intravenous infusion, Day 1, Q3W. Duration: Continuous administration until disease progression, death, intolerable toxicity, subject's voluntary withdrawal, investigator's decision for withdrawal, or a maximum of 24 months.
Radiation: Radiotherapy — Site Selection: Original site, lymph nodes, lung metastasis, bone metastasis, adrenal metastasis, brain metastasis, and other relatively isolated, well-vascularized lesions. Select at least one suitable lesion for radiotherapy based on the impact of the recurrent or metastatic lesion on the body, prioritizing lesions that cause symptoms, are life-threatening, or are expected to cause symptoms.All tumor lesions will be irradiated, which can be done in phases. Dosage and Fractionation: Conventional or hypofractionated radiotherapy, with a biologically effective dose (BED) of ≥ 72 Gy. Dose adjustments can be made for brain metastases. Timing: After completing relevant baseline examinations, radiotherapy can be implemented generally after 4-6 cycles of systemic therapy, or after the first cycle for small, solitary metastatic lesions. echnique: IMRT, TOMO, SBRT, 3D-BT, interstitial implantation therapy, or proton therapy.

SUMMARY:
The goal of this clinical trial is to evaluation the efficacy and safety of iparomlimab and tuvonralimab, paclitaxel + cisplatin/carboplatin combined with radiotherapy of locally recurrent and oligometastatic cervical cancer.The main questions it aims to answer are:

1. Does the combination therapy improve the overall response rate (ORR), progression-free survival (PFS), disease control rate (DCR), overall survival (OS), and safety in participants?
2. What are the predictive biomarkers of treatment efficacy, and how can this information better guide the use of immune-oncology drugs in combination therapy?

Participants will:

* Receive iparomlimab and tuvonralimab, Paclitaxel + Cisplatin/Carboplatin and radiation therapy according to a specified protocol.
* Visit the clinic for regular checkups and tests throughout the treatment period.
* Be monitored for and have records kept of ORR, PFS, DCR, OS, and safety.
* Provide hematologic、tissue and stool samples to explore biomarkers.

This study will help determine if this combination therapy can become a new standard of care for patients with locally recurrent and oligometastatic cervical cancer as well as identify biomarkers to better guide treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to any trial-related procedures;
2. Female, aged ≥18 and ≤75 years;
3. ECOG PS 0-1;
4. Histologically or cytologically confirmed primary cervical cancer (squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma) at initial diagnosis, meeting clinical diagnostic criteria;
5. Locally recurrent or oligometastatic cervical cancer after initial treatment. Total recurrent + metastatic lesions ≤5.Oligometastasis criteria:Lymph node metastases within the same region = 1 lesion;Liver metastases ≤1 lesion;Lung metastases ≤3 lesions
6. At least one measurable lesion (including primary lesion) suitable for radiotherapy and evaluable per RECIST v1.1;
7. Available tumor tissue sample for biomarker assessment;
8. Expected survival ≥6 months;
9. Normal organ function (within 7 days pre-enrollment):

(1) Hematological criteria (no transfusion/granulocyte/platelet-stimulating drugs within 14 days):

1. Hemoglobin (Hb) ≥80 g/L
2. Absolute neutrophil count (ANC) ≥1.5×10⁹/L
3. Platelets (PLT) ≥50×10⁹/L (2) No functional organic disease:

a) ALT/AST ≤2.5×ULN, total bilirubin ≤1.5×ULN, ALP ≤3×ULN, albumin ≥30 g/L b) Serum Cr ≤1.5×ULN (if >1.5×ULN, CrCl ≥50 mL/min by Cockcroft-Gault formula) c) PT prolongation ≤6 sec, APTT ≤1.5×ULN d) TSH ≤ULN (if abnormal, FT3/FT4 must be normal) f) LVEF >50% 10. Prior anti-tumor treatment toxicities recovered to ≤Grade 1 (CTCAE v5.0) pre-treatment, excluding:

* Alopecia/pigmentation (any grade)
* Peripheral neuropathy (≤Grade 2)
* Other toxicities where benefit-risk favors treatment 11. Non-sterilized/childbearing-potential females must:
* Use medical contraception (IUD/oral contraceptives/condoms) during treatment + 3 months post-treatment
* Negative serum/urine HCG within 7 days pre-enrollment
* Non-lactating 12. Expected compliance with protocol follow-up following criteria:

  1. Prior immunotherapy (e.g., immune checkpoint inhibitors);
  2. Pathological diagnosis of gastric-type adenocarcinoma;
  3. Active autoimmune disease or history of autoimmune disease (including but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, hypothyroidism). Exceptions: vitiligo; childhood asthma fully resolved without intervention in adulthood. Exclusion: asthma requiring bronchodilator therapy;
  4. Current use of immunosuppressants or systemic/absorbable topical corticosteroids (equivalent to >10 mg/day prednisone) for immunosuppression, continued within 2 weeks before enrollment;
  5. History of Grade 3-4 immune-related adverse events (irAEs) associated with prior anti-tumor immunotherapy;
  6. Poorly controlled cardiac conditions:

  <!-- -->

  1. NYHA Class II or higher heart failure
  2. Unstable angina
  3. Myocardial infarction within 6 months
  4. Clinically significant supraventricular/ventricular arrhythmia requiring treatment
  5. QTc >450 ms (males) or >470 ms (females); 7. Coagulation abnormalities (INR >1.5 or PT >16 s), bleeding tendency, or current thrombolytic/anticoagulant therapy; 8. Prior radiotherapy/chemotherapy/hormonal therapy/surgery/targeted therapy completed <4 weeks before study treatment (or <5 drug half-lives, whichever is longer); unresolved toxicities (excluding alopecia) from prior therapies >CTCAE Grade 1; 9. Poorly controlled third-space effusion requiring drainage before first trial drug administration; 10. Significant hemoptysis (≥2.5 mL/day) within 2 months before randomization; 11. Known hereditary/acquired bleeding/thrombotic disorders (e.g., hemophilia, coagulation dysfunction, thrombocytopenia, hypersplenism); 12. Active infection or unexplained fever >38.5°C during screening/before first dose; 13. Objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-induced pneumonitis, or severe pulmonary dysfunction; 14. Immunodeficiency (e.g., HIV infection) or active hepatitis:

     * HBV DNA > upper limit of normal (ULN)
     * HCV RNA > ULN; 15. Use of other investigational drugs within 4 weeks before first dose; radiotherapy/local therapy within 2 weeks without full recovery; 16. Concurrent/prior malignancies (except cured basal cell carcinoma/cervical carcinoma in situ); 17. Planned concurrent systemic anti-tumor therapy during the study; 18. Live vaccination within 4 weeks before treatment or planned during the study; 19. Other conditions potentially requiring study termination per investigator judgment:
     * Severe comorbidities (including psychiatric disorders) requiring treatment
     * Critical lab abnormalities
     * Social/family factors compromising safety or data/sample collection.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | Progression-Free Survival (PFS) will be assessed from the date of enrollment until the date of first documented disease progression or death from any cause, whichever occurs first, assessed up to 60 months
  Progression-Free Survival (PFS) will be assessed from the date of enrollment until the date of first documented disease progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate | Assessed every 6 weeks via imaging until study completion (up to 24 months
  ORR refers to the proportion of patients whose optimal response is complete or partial response
Overall Survival | The time interval from enrollment to death from any cause, assessed up to 60 months
  The time interval from enrollment to death from any cause
Disease Control Rate | Assessed every 6 weeks via imaging until study completion (up to 24 months）
  DCR refers to the proportion of patients whose optimal response is complete or partial response, or stable disease
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | Before each chemotherapy cycle (each cycle is 21 days), at 24 hours pre- and post-radiotherapy, and every 3 months during follow-up (up to 24 months)
  Number of participants with adverse events and severe as assessed by CTCAE v5.

CONTACTS AND LOCATIONS:
Overall Officials: Peng Xie, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital Affiliated to Shandong First Medical University, Jinan, Shandong Recruiting, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol